CLINICAL TRIAL: NCT01010542
Title: A SINGLE DOSE STUDY OF THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS AND CLINICAL ACTIVITY OF ILV-095 ADMINISTERED SUBCUTANEOUSLY TO SUBJECTS WITH PSORIASIS.
Brief Title: Study Evaluating Single Dose Of ILV-095 In Psoriasis Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 3226K1-1002; B1991002 (Other: Alias Study Number)
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Plaque Psoriasis
Keywords: Single dose psoriasis study

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ILV-095 (Active Comparator)
  Interventions: Drug: ILV-095 300 mg in a 4 to 1 ratio
- placebo (Placebo Comparator)
  Interventions: Drug: ILV-095 300 mg in a 4 to 1 ratio

INTERVENTIONS:
Drug: ILV-095 300 mg in a 4 to 1 ratio — Single dose of ILV-095 300 mg
  Arms: ILV-095
Drug: ILV-095 300 mg in a 4 to 1 ratio — Single dose of Placebo
  Arms: placebo

SUMMARY:
The purpose of this research study is to evaluate the safety and tolerability of ILV-095 when it is given to individuals with moderate to severe chronic plaque psoriasis. Another purpose of the study is to observe how the drug enters the blood and tissues over time, how the body breaks down the drug and whether or not the body will develop an immune reaction (sensitivity) to the drug.

DETAILED DESCRIPTION:
B1991002 study is a phase 1 adaptive design study which terminated on 14Mar2011. Regular analyzes of psoriasis assessments conducted per the statistical plan indicate that even if every patient enrolled for the rest of the study respond (up to 23 additional subjects), the study can not meet its primary efficacy endpoint. Pfizer Inc. has terminated the trial and clinical team is asking all clinical investigators to continue collecting safety, pharmacokinetics and pharmacodynamics data until the last subject last visit for all subjects who received test article. Last Subject Last Visit occurred 20May2011.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active men or women must agree to use a medically acceptable form of contraception during the study and continue it for 16 weeks after investigational product administration.
* Negative urine pregnancy test result for all women.
* Body mass index (BMI) >=18 kg/m2 and body weight >=50 kg. BMI is calculated by taking the subject's weight, in kilograms, divided by the square of the subject's height, in meters, at screening: BMI = weight (kg)/(height [m]).
* Must meet the following criteria for disease activity, at screening and/or at study entry (subjects who washout from prior therapy may not meet this level of disease activity at screening but must before being entered into the study).
* Must have stable moderate to severe chronic plaque psoriasis covering >=15% of body surface area and be a candidate for systemic therapy or phototherapy.
* Psoriasis Area Severity Index (PASI) score of >11.
* Physician Global Assessment (PGA) of psoriasis score >=3.
* Target lesion score >=6 based on the physician rating of selected sites for erythema, plaque elevation and scaling, with a minimum of 2 on the plaque elevation score. A-12-point score will be used with a 1-4 scale for each domain. Target lesions should not be on the scalp, axillae, face, or groin.

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Evidence of unstable clinically significant disease (eg, unstable cardiovascular, renal, respiratory, or psychiatric disease or any serious disorder that currently requires physician care).
* Acute disease state (eg, nausea, vomiting, fever, or diarrhea) within 7 days before study day 1.
* Evidence of skin conditions (eg, eczema) other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis.
* Presence of guttate, erythrodermic, or pustular psoriasis.
* Active severe infections within 4 weeks before study day 1.
* Systemic malignancy within the past 5 years including melanoma. Treated skin cancer (basal cell carcinoma or squamous cell carcinoma) is excluded.

Evidence of latent tuberculosis by purified protein derivative (PPD) screening. PPD screening should be performed according to local standards using the tuberculin skin test (TST). Any result >5mm is considered positive. Prior Bacillus Calmette-Guerin (BCG) should not be taken into account when interpreting a TST result. TST must be performed during the screening period unless one has been performed within the previous 3 months and the results are available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2011-05-20 (Actual); Study Completion 2011-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (7):
  - Cetero Research, Miami Gardens, Florida
  - Miami Research Associates, Inc., South Miami, Florida
  - MRA Clinical Research, South Miami, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Radiant Research, Inc., Greer, South Carolina
- Canada (2):
  - NewLab Clinical Research Inc, St. John's, Newfoundland and Labrador
  - K. Papp Clinical Research, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3226K1-1002&StudyName=Study%20Evaluating%20Single%20Dose%20Of%20ILV-095%20In%20Psoriasis%20Subjects

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was early terminated based on the outcome of interim analysis which was conducted when data from 39 participants was available. At the time of study termination, 30 participants had received 300 milligram (mg) of ILV-095, 8 participants had received placebo, and 1 participant had received 100 mg of ILV-095.
Groups:
- ILV-095 100 mg: Participants received single dose of ILV-095 100 mg subcutaneously on Day 1 and were followed up to Week 16.
- ILV-095 300 mg: Participants received single dose of ILV-095 300 mg subcutaneously on Day 1 and were followed up to Week 16.
- Placebo: Participants received single dose of placebo matching to ILV-095 subcutaneously on Day 1 and were followed up to Week 16.
Period: Overall Study
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Started | 1 | 30 | 8
Completed | 1 | 25 | 6
Not Completed | 0 | 5 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all randomly assigned participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo | Total
Number analyzed (Participants) | 1 | 30 | 8 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.00 (0.00) | 46.23 (12.94) | 44.63 (8.90) | 45.41 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 3 | 9
  Male | 1 | 24 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 50 Percent Improvement From Baseline in Total Psoriasis Area Severity Index (PASI) Score at Week 2
Description: PASI score: combined assessment of lesion severity and area affected into single score range:0 (no disease) to 72(maximal disease),with higher scores representing greater severity of psoriasis.Body divided into 4 sections(head and neck [h],arms [u],trunk [t],legs [l]);each area scored by itself and scores combined for final PASI score.For each section,percent body surface area(A) of skin involved was estimated:0 (no involvement) to 6 (90 to 100 percent involvement),severity estimated by clinical signs:erythema(E),infiltration(I),scaling(S);5 point scale:0(no involvement) to 4(very marked involvement).Final PASI score = 0.1Ah(Eh + Ih + Sh) + 0.2Au(Eu + Iu + Su) + 0.3At(Et + It + St) + 0.4Al(El + Il + Sl),where head:0.1;upper limbs:0.2;trunk:0.3;lower limbs:0.4. Percentage of participants with at least 50 percent(%) improvement in total PASI score at Week 2 relative to baseline total PASI score was reported and 95% confidence interval was calculated using Clopper-Pearson (exact) method.
Time Frame: Baseline, Week 2
Population: Intent-to-treat (ITT) population included all randomly assigned participants who took at least 1 dose of study medication and had at least 1 clinical activity measurement (PASI score). Here, "Number of Participants Analyzed" (N) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 29 | 7
percentage of participants | 0 [0.0 to 97.5] | 13.8 [3.9 to 31.7] | 14.3 [0.4 to 57.9]

2. Primary Outcome: Percentage of Participants With 50 Percent Improvement From Baseline in Total Psoriasis Area Severity Index (PASI) Score at Week 4
Description: PASI score: combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72(maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u],trunk [t],legs [l]);each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated: 0 (no involvement) to 6 (90 to 100 percent involvement),severity estimated by clinical signs: erythema(E),infiltration(I),scaling(S);5 point scale:0(no involvement) to 4(very marked involvement).Final PASI score = 0.1Ah(Eh + Ih + Sh) + 0.2Au(Eu + Iu + Su) + 0.3At(Et + It + St) + 0.4Al(El + Il + Sl),where head:0.1;upper limbs:0.2;trunk:0.3;lower limbs:0.4. Percentage of participants with at least 50% improvement in total PASI score at Week 4 relative to baseline total PASI score was reported and 95% confidence interval was calculated using Clopper-Pearson (exact) method.
Time Frame: Baseline, Week 4
Population: ITT population included all randomly assigned participants who took at least 1 dose of study medication and had at least 1 clinical activity measurement (PASI score). Here, "N" signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 28 | 7
percentage of participants | 0 [0.0 to 97.5] | 28.6 [13.2 to 48.7] | 28.6 [3.7 to 71.0]

3. Primary Outcome: Percentage of Participants With 50 Percent Improvement From Baseline in Total Psoriasis Area Severity Index (PASI) Score at Week 6
Description: PASI score: combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72(maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u],trunk [t],legs [l]);each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated: 0 (no involvement) to 6 (90 to 100 percent involvement),severity estimated by clinical signs: erythema(E),infiltration(I),scaling(S);5 point scale:0(no involvement) to 4(very marked involvement).Final PASI score = 0.1Ah(Eh + Ih + Sh) + 0.2Au(Eu + Iu + Su) + 0.3At(Et + It + St) + 0.4Al(El + Il + Sl),where head:0.1;upper limbs:0.2;trunk:0.3;lower limbs:0.4. Percentage of participants with at least 50% improvement in total PASI score at Week 6 relative to baseline total PASI score was reported and 95% confidence interval was calculated using Clopper-Pearson (exact) method.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 28 | 6
percentage of participants | 0 [0.0 to 97.5] | 25.0 [10.7 to 44.9] | 33.3 [4.3 to 77.7]

4. Primary Outcome: Percentage of Participants With 50 Percent Improvement From Baseline in Total Psoriasis Area Severity Index (PASI) Score at Week 8
Description: PASI score: combined assessment of lesion severity and area affected into single score range: 0 (no disease) to 72(maximal disease), with higher scores representing greater severity of psoriasis. Body divided into 4 sections (head and neck [h], arms [u],trunk [t],legs [l]);each area scored by itself and scores combined for final PASI score. For each section, percent body surface area (A) of skin involved was estimated: 0 (no involvement) to 6 (90 to 100 percent involvement),severity estimated by clinical signs: erythema(E),infiltration(I),scaling(S);5 point scale:0(no involvement) to 4(very marked involvement).Final PASI score = 0.1Ah(Eh + Ih + Sh) + 0.2Au(Eu + Iu + Su) + 0.3At(Et + It + St) + 0.4Al(El + Il + Sl),where head:0.1;upper limbs:0.2;trunk:0.3;lower limbs:0.4. Percentage of participants with at least 50% improvement in total PASI score at Week 8 relative to baseline total PASI score was reported and 95% confidence interval was calculated using Clopper-Pearson (exact) method.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 27 | 6
percentage of participants | 0 [0.0 to 97.5] | 33.3 [16.5 to 54.0] | 16.7 [0.4 to 64.1]

5. Other Pre Specified Outcome: Target Lesion Score (TLS)
Description: Each lesion was evaluated for 3 components: erythema, plaque elevation, and scaling. Physician rated each component using the following scale: 0= none, 1= mild, 2= moderate, 3= severe and 4= very severe, where higher scores indicated higher lesion severity. TLS was calculated as the sum of the 3 individual components and TLS total score ranged from 0 (no disease) to 12 (maximal disease severity), where higher scores indicated more severity.
Time Frame: Pre-treatment (Day -1), Week 2, 4, 6, 8
Population: ITT population included all randomly assigned participants who took at least 1 dose of study medication and had at least 1 clinical activity measurement (PASI score). Here, "n" signifies those participants who were evaluable for this measure at specified time-points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
units on a scale
  Day -1 | 9.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 7.77 (1.41) | 8.13 (0.83)
  Week 2: number analyzed (Participants) | 1 | 29 | 8
  Week 2 | 8.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 5.93 (2.33) | 6.63 (2.26)
  Week 4: number analyzed (Participants) | 1 | 28 | 8
  Week 4 | 6.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 5.11 (2.60) | 4.75 (2.87)
  Week 6: number analyzed (Participants) | 1 | 28 | 7
  Week 6 | 6.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 4.64 (3.02) | 4.43 (2.88)
  Week 8: number analyzed (Participants) | 1 | 27 | 7
  Week 8 | 4.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 4.63 (3.05) | 5.29 (2.98)

6. Other Pre Specified Outcome: Physician Global Assessment (PGA) Score of Psoriasis
Description: PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema (E), infiltration (I), and scaling (S) across all psoriatic lesions. The severity rating scores (erythema: 0= no evidence of erythema to 4= dark, deep red; infiltration: 0= no evidence of plaque elevation to 4= marked plaque elevation, hard/sharp borders; scaling: 0= no evidence of scaling to 4= thick, coarse scale predominates) were summed (E + I + S = total) and the average (total score divided by 3) was calculated. The average was rounded to the nearest whole number score to determine the PGA. The 5-point scale for PGA was ranging from: 0= clear; 1= almost clear; 2= mild; 3= moderate; 4= severe, where higher scores indicated more severity.
Time Frame: Pre-treatment (Day -1), Week 2, 4, 6, 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
units on a scale
  Day -1 | 4.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 3.23 (0.43) | 3.38 (0.52)
  Week 2: number analyzed (Participants) | 1 | 29 | 8
  Week 2 | 3.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 2.52 (0.87) | 3.00 (0.76)
  Week 4: number analyzed (Participants) | 1 | 28 | 8
  Week 4 | 3.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 2.25 (0.97) | 2.63 (0.92)
  Week 6: number analyzed (Participants) | 1 | 28 | 7
  Week 6 | 3.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 2.18 (0.98) | 2.86 (0.69)
  Week 8: number analyzed (Participants) | 1 | 27 | 7
  Week 8 | 3.00 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 2.37 (1.01) | 2.71 (0.76)

7. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities of Potential Clinical Importance
Description: Hematology (decrease of greater than or equal to [>=] 5% hematocrit, hemoglobin >=20 gram per liter [g/L]; white blood cell less than [<] 3.0*10^9/L; neutrophil <1.5*10^9/L; platelet <100*10^9 /L; eosinophil greater than [>] 0.5*10^9/L); coagulation (prothrombin, partial thromboplastin time >1.5*upper limit of normal [ULN]); chemistry (above ULN or below lower limit of normal [LLN] for [sodium >5 millimole per liter {mmol/L}; potassium >0.5 mmol/L; glucose {fasting} >0.83 mmol/L; glucose {non fasting} >5.0 mmol/L; phosphorus >0.162 mmol/L]; creatinine >1.36*ULN; blood urea nitrogen/urea >1.5*ULN; creatine kinase >3*ULN; change from baseline in [calcium >=0.25 mmol/L; magnesium >=0.21 mmol/L; total protein >=20 g/L; albumin >=10 g/L; uric acid >0.119 mmol/L]; fasting [cholesterol >7.77 mmol/L; triglyceride >3.39 mmol/L]); liver test (alanine amino [A] transferase [T], aspartate AT, total bilirubin >2*ULN; alkaline phosphatase >1.5*ULN; gamma glutamyl T, lactate dehydrogenase >3*ULN).
Time Frame: Baseline (Day 1) up to Week 16
Population: Safety population included all randomly assigned participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
participants | 1 | 19 | 6

8. Other Pre Specified Outcome: Number of Participants With Vital Sign Abnormalities of Potential Clinical Importance
Description: Sitting and supine systolic blood pressure (BP): increase of >=20 millimeter mercury (mm Hg) from baseline value and >=160 mm Hg; decrease of >=20 mm Hg from baseline value and less than or equal to (<=) 90 mm Hg. Diastolic BP: increase of >=15 mm Hg from baseline value and >=100 mm Hg; decrease of >=15 mm Hg from baseline value and <=50 mm Hg. Heart rate: increase of >15 beats per minute (bpm) from baseline value and >=120 bpm; decrease of >15 bpm from baseline value and <=45 bpm. Orthostatic (supine to standing): 1) systolic BP: decrease of >=20 mm Hg from supine value; 2) diastolic BP: decrease of >=20 mm Hg from supine value; 3) heart rate: increase of >=30 bpm from supine value. Oral temperature <35 degree Celsius or >38.3 degree Celsius. Respiratory rate <10 breaths per minute; >25 breaths per minute. Weight >=7% increase or decrease from baseline value.
Time Frame: Baseline (Day 1) up to Week 16
Population: Safety population included all randomly assigned participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
participants | 0 | 6 | 2

9. Other Pre Specified Outcome: Number of Participants With Electrocardiograms (ECG) Abnormalities of Potential Clinical Importance
Description: Criteria for abnormality of potential clinical importance: PR interval: change of >=20 milliseconds (msec) from baseline value and >=220 msec; QRS interval: >=120 msec; corrected QT (QTc) interval (men): >450 msec and QTc interval (women): >470 msec.
Time Frame: Baseline (Day 1) up to Week 16
Population: Safety population included all randomly assigned participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
participants | 1 | 24 | 8

10. Other Pre Specified Outcome: Maximum Observed Serum Concentration (Cmax) of ILV-095
Time Frame: Pre-dose, 2, 4, 8, 24, 48, 120, 216, 312, 480, 648, 984, 1320, 1656, 1992, 2328, 2664 hours post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomly assigned participants who took at least 1 dose of ILV-095 and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | ILV-095 100 mg | ILV-095 300 mg
Number analyzed (Participants) | 1 | 30
microgram per milliliter (mcg/mL) | 7.39 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 19.25 (8.1558)

11. Other Pre Specified Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of ILV-095
Time Frame: Pre-dose, 2, 4, 8, 24, 48, 120, 216, 312, 480, 648, 984, 1320, 1656, 1992, 2328, 2664 hours post-dose
Population: PK parameter analysis population included all randomly assigned participants who took at least 1 dose of ILV-095 and had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: days
Arm/Group | ILV-095 100 mg | ILV-095 300 mg
Number analyzed (Participants) | 1 | 30
days | 2.01 [NA to NA] — Full range could not be estimated as only 1 participant was analyzed. | 5.98 [1.97 to 9.21]

12. Other Pre Specified Outcome: Serum Terminal Half-Life (t1/2) of ILV-095
Description: t1/2 was the time measured for the serum concentration of ILV-095 to decrease by one half.
Time Frame: Pre-dose, 2, 4, 8, 24, 48, 120, 216, 312, 480, 648, 984, 1320, 1656, 1992, 2328, 2664 hours post-dose
Population: PK parameter analysis population included all randomly assigned participants who took at least 1 dose of ILV-095 and had at least 1 of the PK parameters of interest. Here, "N" signifies number of participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ILV-095 100 mg | ILV-095 300 mg
Number analyzed (Participants) | 1 | 29
days | 13.0 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 15.40 (2.7272)

13. Other Pre Specified Outcome: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of ILV-095
Description: AUCinf was calculated as AUClast + (Clast/kel), where AUClast was area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (Clast) and Kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose, 2, 4, 8, 24, 48, 120, 216, 312, 480, 648, 984, 1320, 1656, 1992, 2328, 2664 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Standard Deviation); unit: microgram*hour per milliliter
Arm/Group | ILV-095 100 mg | ILV-095 300 mg
Number analyzed (Participants) | 1 | 28
microgram*hour per milliliter | 5070 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 13200 (6828.5)

14. Other Pre Specified Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Time of The Last Quantifiable Concentration (AUClast) of ILV-095
Description: AUClast was the area under the serum concentration versus time curve from time zero to the time of the last quantifiable concentration (Clast).
Time Frame: Pre-dose, 2, 4, 8, 24, 48, 120, 216, 312, 480, 648, 984, 1320, 1656, 1992, 2328, 2664 hours post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: microgram*hour per milliliter
Arm/Group | ILV-095 100 mg | ILV-095 300 mg
Number analyzed (Participants) | 1 | 30
microgram*hour per milliliter | 5040 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 12190 (6803.3)

15. Other Pre Specified Outcome: Apparent Clearance (CL/F) of ILV-095
Description: Clearance was a quantitative measure of the rate at which ILV-095 was removed from the blood (rate at which ILV-095 was metabolized or eliminated by normal biological processes).
Time Frame: Pre-dose, 2, 4, 8, 24, 48, 120, 216, 312, 480, 648, 984, 1320, 1656, 1992, 2328, 2664 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | ILV-095 100 mg | ILV-095 300 mg
Number analyzed (Participants) | 1 | 28
liter per hour (L/hr) | 0.0197 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 0.02275 (0.022558)

16. Other Pre Specified Outcome: Apparent Volume of Distribution (Vz/F) of ILV-095
Description: Apparent volume of distribution was defined as the theoretical volume in which the total amount of ILV-095 was needed to be uniformly distributed to produce the desired serum concentration of ILV-095.
Time Frame: Pre-dose, 2, 4, 8, 24, 48, 120, 216, 312, 480, 648, 984, 1320, 1656, 1992, 2328, 2664 hours post-dose
Population: as for outcome 12
Measure: Geometric Mean (Standard Deviation); unit: liter
Arm/Group | ILV-095 100 mg | ILV-095 300 mg
Number analyzed (Participants) | 1 | 28
liter | 8.90 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 11.83 (10.656)

17. Other Pre Specified Outcome: Serum Amyloid-A Levels
Description: Serum amyloid-A (SAA) is a low molecular weight acute phase protein. Serum samples were analyzed for SAA concentrations using solid phase sandwich enzyme-linked immunosorbent assay. The limit of detection (LOD) for SAA assay was 0.21 ng/mL.
Time Frame: Baseline, Day 14, 56,112
Population: Safety population included all randomly assigned participants who took at least 1 dose of study medication. Here, "n" signifies those participants who were evaluable for this measure at specified time-points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
nanogram per milliliter (ng/mL)
  Baseline | 53753.0 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 53161.8 (86984.7) | 24316.5 (14098.6)
  Day 14: number analyzed (Participants) | 1 | 29 | 8
  Day 14 | 74142.0 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 64341.8 (121231.2) | 27118.9 (14287.6)
  Day 56: number analyzed (Participants) | 1 | 27 | 7
  Day 56 | 114900.0 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 45934.9 (62741.2) | 40405.6 (55721.3)
  Day 112: number analyzed (Participants) | 1 | 29 | 8
  Day 112 | 62092.0 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 38173.3 (29227.6) | 25537.1 (9639.5)

18. Other Pre Specified Outcome: Plasma Interleukin-6 (IL-6) Levels
Description: Interleukin: group of naturally occurring proteins that are particularly important in stimulating immune responses such as inflammation. Plasma samples were analyzed for IL-6 concentrations using high sensitive enzyme-linked immunosorbent assay. The limit of detection for IL-6 assay was 0.00002 ng/mL.
Time Frame: Baseline, Day 14, 56,112
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 2 | 60 | 16
nanogram per liter (ng/L)
  Baseline | 4.7 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 4.8 (7.6) | 3.6 (2.4)
  Day 14: number analyzed (Participants) | 2 | 58 | 16
  Day 14 | 6.0 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 5.5 (6.8) | 3.4 (2.6)
  Day 56: number analyzed (Participants) | 2 | 54 | 14
  Day 56 | 4.7 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 4.8 (5.5) | 2.9 (1.3)
  Day 112: number analyzed (Participants) | 2 | 58 | 15
  Day 112 | 5.4 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 4.5 (4.4) | 2.6 (1.5)

19. Other Pre Specified Outcome: Plasma Interleukin-22 (IL-22) Levels
Description: Interleukin: group of naturally occurring proteins that are particularly important in stimulating immune responses such as inflammation. Plasma samples were analyzed for IL-22 concentrations using highly sensitive enzyme-linked immunosorbent assay. The lower limit of quantification for IL-22 assay was 0.34 pg/mL.
Time Frame: Baseline, Day 14, 56,112
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
picogram per milliliter (pg/mL)
  Baseline | 636.9 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 334.4 (352.7) | 1150.4 (1229.3)
  Day 14: number analyzed (Participants) | 1 | 29 | 8
  Day 14 | 5688.3 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 1273.9 (1642.4) | 733.3 (708.4)
  Day 56: number analyzed (Participants) | 1 | 27 | 7
  Day 56 | 7412.3 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 2886.6 (2260.5) | 552.0 (377.5)
  Day 112: number analyzed (Participants) | 1 | 27 | 8
  Day 112 | 2202.4 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 3471.3 (2368.0) | 363.1 (273.6)

20. Other Pre Specified Outcome: Serum C-Reactive Protein (CRP) Levels
Description: CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation. Serum samples were analyzed for CRP concentrations using nephelometry.
Time Frame: Baseline, Day 14, 56,112
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
milligram per liter (mg/L)
  Baseline | 11.2 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 7.2 (6.7) | 4.7 (1.9)
  Day 14: number analyzed (Participants) | 1 | 29 | 8
  Day 14 | 9.6 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 9.1 (10.9) | 5.0 (1.9)
  Day 56: number analyzed (Participants) | 1 | 27 | 6
  Day 56 | 13.0 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 6.4 (6.7) | 4.9 (2.2)
  Day 112: number analyzed (Participants) | 1 | 28 | 8
  Day 112 | 12.1 (NA) — Standard deviation could not be estimated as only 1 participant was analyzed. | 6.1 (3.2) | 4.6 (1.8)

21. Other Pre Specified Outcome: Number of Participants With Positive Anti-Drug Antibodies of ILV-095
Description: The serum samples were analyzed for anti-drug antibodies of ILV-095 by a validated electrochemiluminescence assay and participants with positive anti-drug antibodies were reported in this outcome measure.
Time Frame: Baseline up to Week 16
Population: Safety population included all randomly assigned participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
participants | 0 | 16 | 0

22. Other Pre Specified Outcome: Number of Participants With Injection-Site Reactions
Description: Injection site reactions included following symptoms: injection site itching, injection site redness, injection-site swelling, injection site pain, injection site ulceration, requirement for plastic surgery associated with an injection.
Time Frame: Baseline up to Week 16
Population: Safety population included all randomly assigned participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Number analyzed (Participants) | 1 | 30 | 8
participants | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | ILV-095 100 mg | ILV-095 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/30 | 0/8
Other Adverse Events (participants affected / at risk) | 0/1 | 22/30 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ILV-095 100 mg (N=1) | ILV-095 300 mg (N=30) | Placebo (N=8)
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ILV-095 100 mg (N=1) | ILV-095 300 mg (N=30) | Placebo (N=8)
Cardiac Failure (Cardiac disorders) | 0 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0
Mydriasis (Eye disorders) | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0
Parotid Gland Inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0
Irritability (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Temperature Intolerance (General disorders) | 0 | 1 | 0
Seasonal Allergy (Immune system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 5 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 1
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 2 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine Aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate Aminotransferase increased (Investigations) | 0 | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 0
C-Reactive Protein Increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1
Impatience (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0
Tension (Psychiatric disorders) | 0 | 1 | 0
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was early terminated based on the outcome of interim analysis and not due to any safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.